CLINICAL TRIAL: NCT06842836
Title: Evaluation of Alterations in the Gut Microbiota in Bronchial Asthma: a Feasibility Study in a Pediatric Population in the Alexandria Area.
Brief Title: Evaluation of Alterations in the Gut Microbiota in Pediatric Bronchial Asthma
Acronym: MicroAsm
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: ASO.Ped.23.11
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Asthma Bronchiale
Keywords: microbiota

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study cohort: Pediatric subjects aged 6 to 9 years, diagnosed with intermittent or mild persistent bronchial asthma, referred to the pediatric outpatient clinic of the Children's Hospital of Alessandria will be enrolled in the study
  Interventions: Other: Study intervention

INTERVENTIONS:
Other: Study intervention — From the date of study authorization, the principal investigator, together with his specially identified collaborators, will proceed to identify patients who meet the inclusion criteria. Then, during the first follow-up visit, the principal investigator, or one of his co-investigators, will deliver the informed consent to the parent(s) of the minor subject candidate for enrollment in the study, explaining all the characteristics and evaluations stipulated in the protocol and answering any questions. After the informed consent is signed, patients will be enrolled and the data required to conduct the study will be collected, and a fecal sample will be requested specifically for the conduct of the study. At the same time, completion of the KIDMED (Mediterranean Diet Quality Index in children and adolescents) questionnaire will be requested.

SUMMARY:
Asthma constitutes a major chronic noncommunicable disease, globally it affects about 300 million people and the incidence has been steadily increasing in recent decades; it affects about 10% of children and is the leading chronic disease in childhood. The microbiota constitutes the collection of all microorganisms-bacteria, viruses, fungi, protozoa-that live in symbiosis with our bodies. Disruption of the microbiota during this critical period of development can cause asthma, allergies, and other immunological disorders. Therefore, it can be an important environmental factor that determines the transition of health to disease. The aim of the intended study is to evaluate and analyze the presence of possible alterations in the gut microbiota in a cohort of pediatric asthmatic subjects by collecting fecal samples.

DETAILED DESCRIPTION:
Asthma constitutes a major chronic noncommunicable disease, globally affecting about 300 million people and the incidence has been steadily increasing in recent decades; it affects about 10% of children and is the leading chronic disease in childhood. Symptoms mainly include airway narrowing and inflammation, which appear to originate from a synergy of environmental and genetic factors. The pathogenesis of asthma is not yet well understood, but it could be related during childhood to several factors such as: antibiotic use during the neonatal period, type of delivery, maternal diet, and formula feeding. It is confirmed that changes in the gut microbiota determine susceptibility to the development of asthma, especially when they occur in the early years of life. The microbiota constitutes the set of all microorganisms-bacteria, viruses, fungi, protozoa-that live in symbiosis with our bodies. Disruption of the microbiota during this critical period of development can cause asthma, allergies, and other immunological disorders. Therefore, it can be an important environmental factor that determines the transition of health to disease. The intestinal microbiota of children is mainly characterized by the presence of species such as Bifidobacterium spp., Faecalibacterium spp., and members of the Lachnospiraceae compared to the adult microbiota, which is more characterized by the presence of species such as Bacteorides spp. Several studies have shown that a dysbiosis of the gut microbiota early in the life course may be related to an increased risk of developing bronchial asthma as age progresses. The natural diversity of the microbiota could also be affected by a range of medications, such as antibiotics, corticosteroids, and antacids. Antibiotics significantly affect the composition of the gut microbiota with immediate and prolonged effect. The aim of the intended study is to assess and analyze the presence of possible alterations in the intestinal microbiota in a cohort of pediatric asthmatic subjects through the collection of fecal samples, which will be analyzed using an iSeq sequencing method at the SC Microbiology and Virology laboratory of the Azienda Ospedaliero Universitaria SS. Antonio e Biagio e C. Arrigo of Alessandria.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent by Parents;
* Age between 6 and 9 years;
* Confirmed diagnosis of bronchial asthma at Alessandria Children's Hospital through spirometry investigation;
* Bronchial asthma classified as intermittent or mild persistent;
* Patients followed at the outpatient clinics of the SC Pediatrics of AOU SS Antonio e Biagio and C. Arrigo of Alessandria.

Exclusion Criteria:

* Taking prolonged systemic therapy for the treatment of bronchial asthma;
* Bronchial asthma classified as moderate persistent or severe persistent;
* Insurmountable language barrier.
* Ongoing antibiotic intake.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Approximately 25 pediatric subjects aged 6 to 9 years, diagnosed with intermittent or mild persistent bronchial asthma, referred to the pediatric outpatient clinic of the Children's Hospital of Alexandria will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative changes in the gut microbiota | Baseline
  The gut microbiota will be analyzed from a fecal sample using the 16S ribosomal RNA gene as the target of hypervariable regions V3-V6 (QIAamp® PowerFecal® Pro DNA Kit Qiagen, Germany) and using the Illumina® iSeq-100 platform for NGS sequencing.

SECONDARY OUTCOMES:
Quantitative characterization of microbial species of gut microbiota | Baseline
  The gut microbiota will be analyzed from fecal sample using the 16S ribosomal RNA gene as the target of hypervariable regions V3-V6 (QIAamp® PowerFecal® Pro DNA Kit Qiagen, Germany) and using the Illumina® iSeq-100 platform for NGS sequencing.
Mediterranean Diet Quality Index in children and adolescents | Baseline
  Score from 0 to 12 points to assess the association between alterations found in the gut microbiota and quality of life in pediatric and adolescent patients.
  A score below 3 points is classified as representative of low adherence to the Mediterranean Diet, a score between 4-7 points as representative of medium adherence to the Mediterranean Diet, while a score above 8 points as representative of high adherence to the Mediterranean Diet.

CONTACTS AND LOCATIONS:
Locations (1):
- SSD Laboratori di Ricerca (DAIRI) - AOU Alessandria, Alessandria, Italy

IPD SHARING:
Plan to Share IPD: No